CLINICAL TRIAL: NCT02186912
Title: A Clinical Evaluation of All-On-4® Treatment Concept in the Mandible or Maxilla on 4 NobelActive®Implants With a Fixed NobelProcera® Implant Bridge
Brief Title: All-On-4® Treatment Concept
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stopped as the performance of the study showed insufficient patient recruitment.
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-185
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Edentulous
Keywords: edentulous; Nobel Active; Nobel Procera; IBO; CAD/CAM
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mandible (Experimental): Nobel Active Nobel Procera IBO
  Interventions: Device: Nobel Active, Nobel Procera IBO
- maxilla (Experimental): Nobel Active Nobel Procera IBO
  Interventions: Device: Nobel Active, Nobel Procera IBO

INTERVENTIONS:
Device: Nobel Active, Nobel Procera IBO
  Other Names: Nobel Active implants; Implant bar

SUMMARY:
Indication : edentulous patients To evaluate and compare the marginal bone level change around tilted and straight NobelActive implants placed in healed sites with All-on-4-treatment concept after immediate function supporting NobelProcera Implant Bridge (fixed) in the mandible and maxilla.

ELIGIBILITY:
The subject is at least 18 years of age (or age of consent) and has passed secession of growth

Obtained informed consent from the subject

Edentulous mandible or maxilla providing sufficient bone whereas a fixed NobelProceraTM Implant bridge on four (4) implants is regarded as an appropriate treatment solution

The subject has an osseous architecture enough to receive four implants and a sufficient amount of bone for placing in healed sites implants with a length of at least 8 mm

The implant site is free from infection and extraction remnants Implants will be placed in healed sites.

Good gingival / periodontal / peri-apical status of opposing teeth/implants

The subject fulfills the prerequisite that a harmonic, stable occlusal relationship can be achieved with opposing natural teeth resp. fixed or removable opposing dentition (tooth or implant based

The subjects as well as the implant site(s) fulfill the criteria for immediate loading.

The subject is in such a physical and mental condition that a 5-year follow-up period can be carried out without foreseeable problems The subject is available for the 5-year term of the investigation

Exclusion Criteria:

The subject is not able to give her/his informed consent of participating

Health conditions, which do not permit the surgical (including anesthesia) or restorative procedure

Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or in subject history Any disorders in the planned implant area such as previous tumors, chronic bone disease or previous irradiation in the head/neck area

Alcohol or drug abuse as noted in subject records or in subject history Smoking of >10 cigarettes/day

Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake

Pathologic occlusion, e.g. severe bruxism or other destructive habits

Lack of opposing dentition or unstable occlusion

Ongoing infections, endodontic or periodontal problems in opposing teeth or implants

Subject shows an unacceptable oral hygiene

Subject has allergic or adverse reactions to the restorative material.

Bone augmentation of more than 3mm vertical height performed less than 6 months prior to planned implant placement.

Bis-phosphonate therapy

Implant insertion torque is <35 Ncm or >70 Ncm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
bone level change around tilted and straight implants | yearly up to 5 years

SECONDARY OUTCOMES:
cumulative survival rate (CSR) | yearly up to 5 years

OTHER OUTCOMES:
Quality of Life | yearly up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin Mainz, Mainz, Rhineland-Palatinate, Germany